CLINICAL TRIAL: NCT01683669
Title: Physiological Research on Variable Pressure Support Ventilation in Patients With Acute Acute Lung Injury: Part I and Part II
Brief Title: Effect of Variable PSV in Acute Lung Injury: Part I and Part II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Paolo Pelosi, Full Professor - Chair of Anesthesiology and Intensive Care Medicine. Chief of Intensive Care Medicine, University of Genova
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 91/12
Record Dates: First submitted 2012-08-29; First posted 2012-09-12 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Acute Lung Injury (ALI); Acute Distress Respiratory Syndrome (ARDS)
Keywords: ALI; ARDS; Noisy pressure support ventilation
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Noisy-PSV 1 (Other): different levels of variable pressure support
  Interventions: Other: Noisy-PSV 1
- Noisy-PSV 2 (Other): different levels of variable pressure support
  Interventions: Other: Noisy-PSV 2

INTERVENTIONS:
Other: Noisy-PSV 1 — Noisy-PSV 1: different levels of variable pressure support (PS) will be randomized: a) PS variability equal to 0%, b) PS variability equal to 45%, c) PS variability equal to 90%.
  Arms: Noisy-PSV 1
Other: Noisy-PSV 2 — Noisy-PSV 2 : different levels of variable Pressure Support (PS) will be randomized: a) PS equal to Baseline and variability 0%; b) PS equal to Baseline and variability set in order achieve an increase or decrease of pressure of 5 cmH2O; c) PS equal to Baseline - 5 cmH2O and variability 0%; d) PS equal to Baseline - 5 cmH2O and set in order achieve an increase or decrease of pressure of 5 cmH2O.
  Arms: Noisy-PSV 2

SUMMARY:
Noisy Pressure Support Ventilation (noisy-PSV) would lead to improved lung function, while preserving respiratory muscle unloading. Basically, noisy PSV differs from other assisted mechanical ventilation modes that may also increase the variability of the respiratory pattern (e.g. proportional assist ventilation) by the fact that the variability does not depend on changes in the patient's inspiratory efforts.

The aim of this study is to evaluate the optimal variability for noisy PSV in patients with ALI based on its effects on respiratory mechanics, breathing comfort, gas exchange, and hemodynamics. The investigators hypothesize that noise in pressure support leads to variations in VT that are able to improve lung function and that physiologic variables respond differently to the degree of variability in pressure support

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Intubated/tracheostomized patients in assisted mechanical ventilation
* PaO2/FiO2 100-300, with PEEP ≥ than 5 cmH2O.

Exclusion Criteria:

* Pregnancy
* History of chronic lung disease (COPD)
* Presence of thoracic drainage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Effect on arterial oxygenation in each setting of variability | after 45 minutes of mechanical ventilation with each level of variable pressure support
  The investigators perform an arterial blood gas and oxygenation is evaluated with PaO2/FiO2 ratio

SECONDARY OUTCOMES:
work of breathing | every 9 minutes, up to 45 minutes, of mechanical ventilation in each level of variable pressure support
  work of breathing will be recorded as pressure-time product (PTP) measured on the esophageal pressure curve.
effects on hemodynamic | after 45 minutes of mechanical ventilation with each level of variable pressure support
  the investigator will record blood pressure and cardiac output
effect on arterial carbon dioxide | after 45 minutes of mechanical ventilation with each level of variable pressure support
  The investigators perform an arterial blood gas and arterial carbon dioxide is evaluated with PaCO2.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pelosi, Professor, Study Director — University of Genoa, Italy
Locations (1):
- Intensive Care Medicine Unit - IRCCS San Martino - IST, Genoa, Italy

REFERENCES:
- [Background] Falk DJ, Deruisseau KC, Van Gammeren DL, Deering MA, Kavazis AN, Powers SK. Mechanical ventilation promotes redox status alterations in the diaphragm. J Appl Physiol (1985). 2006 Oct;101(4):1017-24. doi: 10.1152/japplphysiol.00104.2006. Epub 2006 May 4. PMID 16675618
- [Background] Esteban A, Anzueto A, Alia I, Gordo F, Apezteguia C, Palizas F, Cide D, Goldwaser R, Soto L, Bugedo G, Rodrigo C, Pimentel J, Raimondi G, Tobin MJ. How is mechanical ventilation employed in the intensive care unit? An international utilization review. Am J Respir Crit Care Med. 2000 May;161(5):1450-8. doi: 10.1164/ajrccm.161.5.9902018. PMID 10806138
- [Background] Seymour CW, Frazer M, Reilly PM, Fuchs BD. Airway pressure release and biphasic intermittent positive airway pressure ventilation: are they ready for prime time? J Trauma. 2007 May;62(5):1298-308; discussion 1308-9. doi: 10.1097/TA.0b013e31803c562f. PMID 17495742
- [Background] Neumann P, Wrigge H, Zinserling J, Hinz J, Maripuu E, Andersson LG, Putensen C, Hedenstierna G. Spontaneous breathing affects the spatial ventilation and perfusion distribution during mechanical ventilatory support. Crit Care Med. 2005 May;33(5):1090-5. doi: 10.1097/01.ccm.0000163226.34868.0a. PMID 15891341
- [Background] Henzler D, Pelosi P, Bensberg R, Dembinski R, Quintel M, Pielen V, Rossaint R, Kuhlen R. Effects of partial ventilatory support modalities on respiratory function in severe hypoxemic lung injury. Crit Care Med. 2006 Jun;34(6):1738-45. doi: 10.1097/01.CCM.0000218809.49883.54. PMID 16625116
- [Background] Suki B, Alencar AM, Sujeer MK, Lutchen KR, Collins JJ, Andrade JS Jr, Ingenito EP, Zapperi S, Stanley HE. Life-support system benefits from noise. Nature. 1998 May 14;393(6681):127-8. doi: 10.1038/30130. No abstract available. PMID 9603516
- [Background] Arold SP, Suki B, Alencar AM, Lutchen KR, Ingenito EP. Variable ventilation induces endogenous surfactant release in normal guinea pigs. Am J Physiol Lung Cell Mol Physiol. 2003 Aug;285(2):L370-5. doi: 10.1152/ajplung.00036.2003. PMID 12851212
- [Background] Boker A, Graham MR, Walley KR, McManus BM, Girling LG, Walker E, Lefevre GR, Mutch WA. Improved arterial oxygenation with biologically variable or fractal ventilation using low tidal volumes in a porcine model of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2002 Feb 15;165(4):456-62. doi: 10.1164/ajrccm.165.4.2108006. PMID 11850336
- [Background] Mutch WA, Lefevre GR, Cheang MS. Biologic variability in mechanical ventilation in a canine oleic acid lung injury model. Am J Respir Crit Care Med. 2001 Jun;163(7):1756-7. doi: 10.1164/ajrccm.163.7.16372c. No abstract available. PMID 11401900
- [Background] Lefevre GR, Kowalski SE, Girling LG, Thiessen DB, Mutch WA. Improved arterial oxygenation after oleic acid lung injury in the pig using a computer-controlled mechanical ventilator. Am J Respir Crit Care Med. 1996 Nov;154(5):1567-72. doi: 10.1164/ajrccm.154.5.8912782.
- [Background] Mutch WA, Harms S, Lefevre GR, Graham MR, Girling LG, Kowalski SE. Biologically variable ventilation increases arterial oxygenation over that seen with positive end-expiratory pressure alone in a porcine model of acute respiratory distress syndrome. Crit Care Med. 2000 Jul;28(7):2457-64. doi: 10.1097/00003246-200007000-00045. PMID 10921579
- [Background] McMullen MC, Girling LG, Graham MR, Mutch WA. Biologically variable ventilation improves oxygenation and respiratory mechanics during one-lung ventilation. Anesthesiology. 2006 Jul;105(1):91-7. doi: 10.1097/00000542-200607000-00017. PMID 16809999
- [Background] Gama de Abreu M, Spieth PM, Pelosi P, Carvalho AR, Walter C, Schreiber-Ferstl A, Aikele P, Neykova B, Hubler M, Koch T. Noisy pressure support ventilation: a pilot study on a new assisted ventilation mode in experimental lung injury. Crit Care Med. 2008 Mar;36(3):818-27. doi: 10.1097/01.CCM.0000299736.55039.3A. PMID 18431269
- [Background] Spieth PM, Carvalho AR, Guldner A, Pelosi P, Kirichuk O, Koch T, de Abreu MG. Effects of different levels of pressure support variability in experimental lung injury. Anesthesiology. 2009 Feb;110(2):342-50. doi: 10.1097/ALN.0b013e318194d06e. PMID 19194161
- [Background] Brower RG, Lanken PN, MacIntyre N, Matthay MA, Morris A, Ancukiewicz M, Schoenfeld D, Thompson BT; National Heart, Lung, and Blood Institute ARDS Clinical Trials Network. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med. 2004 Jul 22;351(4):327-36. doi: 10.1056/NEJMoa032193. PMID 15269312
- [Derived] Ball L, Sutherasan Y, Fiorito M, Dall'Orto A, Maiello L, Vargas M, Robba C, Brunetti I, D'Antini D, Raimondo P, Huhle R, Schultz MJ, Rocco PRM, Gama de Abreu M, Pelosi P. Effects of Different Levels of Variability and Pressure Support Ventilation on Lung Function in Patients With Mild-Moderate Acute Respiratory Distress Syndrome. Front Physiol. 2021 Oct 22;12:725738. doi: 10.3389/fphys.2021.725738. eCollection 2021. PMID 34744766